CLINICAL TRIAL: NCT05126472
Title: Phase I Study Evaluating the Safety and Tolerability of Locally Administered Anti-CD40 Agonist Antibody (2141-V11) in Subjects With Bladder Cancer
Brief Title: Study of 2141-V11 in People With Non-muscle Invasive Bladder Cancer That Did Not Respond to Standard Treatment
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Pin Down Bladder Cancer Research Foundation (Unknown); Rockefeller University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 21-314
Record Dates: First submitted 2021-11-08; First posted 2021-11-19 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Non-muscle Invasive Bladder Cancer
Keywords: 2141-V11; 21-314
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a phase I, open-label study to assess safety and tolerability of a local delivery (intravesically or intratumorally) of an anti-CD40 agonist antibody (2141-V11) for the treatment of subjects with BCG-unresponsive NMIBC who are considered ineligible for or have elected not to undergo radical cystectomy.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- (Cohort A) anti-CD40 antibody 2141-V11 (Experimental): Intravesically or intratumorally) of an anti-CD40 agonist antibody (2141-V11) for the treatment of subjects with BCG-unresponsive NMIBC who are considered ineligible for or have elected not to undergo radical cystectomy.
  Interventions: Drug: anti-CD40 antibody 2141-V11
- (Cohort B) 2141-V11, a fixed dose of 10mg (Experimental): For patients who are ineligible for radical cystectomy or have elected not to undergo the procedure.
  Interventions: Drug: anti-CD40 antibody 2141-V11
- (Cohort C) expansion cohort 10 mg of 2141-V11 (Experimental): For patients in Cohort C, 10 mg of 2141-V11 will be administered as an intratumoral injection during standard of care cystoscopy prior to and within four weeks of planned radical cystectomy.
  Interventions: Drug: anti-CD40 antibody 2141-V11

INTERVENTIONS:
Drug: anti-CD40 antibody 2141-V11 — Cohort A Eligible subjects will receive the anti-CD40 antibody 2141-V11 administered by intravesical instillation once weekly for 3 consecutive weeks (weeks 1, 2, and 3) for a total of 3 doses. As discussed further below, depending on disease status at week 13 and week 25 evaluations, subjects may be eligible for re-treatment (once weekly for 3 doses) at these time points.
  Arms: (Cohort A) anti-CD40 antibody 2141-V11
Drug: anti-CD40 antibody 2141-V11 — Cohort B Eligible subjects will receive the anti-CD40 antibody 2141-V11 administered by intratumoral injection once every 3 weeks (weeks 1, 4, 7, and 10) for a total of 4 doses. As discussed further below, depending on disease status at week 14 and week 26 evaluations, subjects may be eligible for re-treatment (once every 3 weeks for a total of 4 doses) at these time points.
  Arms: (Cohort B) 2141-V11, a fixed dose of 10mg
Drug: anti-CD40 antibody 2141-V11 — Cohort C Eligible subjects will receive the anti-CD40 antibody 2141-V11 administered by intratumoral injection as a single 10mg during standard of care cystoscopy and examination prior to and within 4 weeks of planned radical cystectomy.
  Arms: (Cohort C) expansion cohort 10 mg of 2141-V11

SUMMARY:
The purpose of this study is to test the safety of the study drug 2141-V11 in people whose NMIBC did not respond to standard treatment, and who will not have the standard surgical procedure to remove the bladder. The researchers will test different doses of 2141-V11 to see which dose is safest in people. The researchers will also do tests to see how the body absorbs, distributes, and gets rid of 2141-V11. This study is one of the first to test 2141-V11 in people, and the first to test 2141-V11 delivered through a catheter into the bladder.

DETAILED DESCRIPTION:
If during Period 1 treatment, the treating physician notices recurrent disease in the bladder, the patient should undergo a biopsy or TURBT. If the pathology returns as HG Ta or CIS, the patient can resume treatment. If pathology returns as HG T1, the patient will be removed from treatment. If a high-grade recurrence occurs during period 2 or 3 treatments, the patient will be removed from treatment.

ELIGIBILITY:
Inclusion Criteria:

Cohorts A and B

* High-grade (HG) NMIBC (HG Ta, CIS, and/or T1) of urothelial histology that is unresponsive to adequate BCG therapy.
* Stage, grade, and histology must be confirmed by the MSK Department of Pathology
* Subjects with tumors of mixed urothelial/non-urothelial histology may be included, but urothelial carcinoma must be the predominant histology; subjects with predominant or exclusively non-urothelial histology are excluded
* In those subjects with CIS, the CIS must be present on the tumor sample from the most recent cystoscopy/TURBT
* In this context, adequate BCG therapy is defined as at least one of the following:
* At least five of six doses of an initial induction course plus at least two of three doses of maintenance therapy
* At least five of six doses of an initial induction course plus at least two of six doses of a second induction course
* Disease unresponsive to adequate BCG therapy is defined as the following. Suspected recurrence from suspicious cytology or cystoscopy, and later confirmed via TURBT, is acceptable:
* Persistent or recurrent CIS alone or with recurrent Ta/T1 disease (noninvasive papillary disease/tumor invades the subepithelial connective tissue) within 12 months of completion of adequate BCG therapy
* Recurrent HG Ta/T1 disease within 6 months of completion of adequate BCG therapy
* HG T1 disease at the first evaluation following an induction BCG course

Cohort C:

* Bladder cancer of any stage that has a predominant urothelial histology.
* Stage, grade, and histology must be confirmed by the MSK Department of Pathology
* Subjects with tumors of mixed urothelial/non-urothelial histology may be included, but urothelial carcinoma must be the predominant histology; subjects with predominant or exclusively non-urothelial histology are excluded

Cohort A and B Only:

* In subjects with papillary tumors (Ta and T1), a complete TURBT must have been performed.

This is characterized by:

* Attainment of a visually complete resection of all papillary tumors (Ta and T1)
* Residual CIS not amenable to complete transurethral resection is acceptable
* Receipt of restaging transurethral resection for any tumor with invasion into the lamina propria (HG T1) as part of standard care, with documented presence of uninvolved detrusor muscle.
* Most recent cystoscopy/TURBT must have been performed within 6 months of the first dose of trial treatment.
* Absence of urothelial carcinoma involving the upper urinary tract (documented by radiological imaging or ureteroscopy).
* Have elected not to undergo or are considered ineligible for radical cystectomy, as determined by the treating surgeon. Reasons for ineligibility or refusal of radical cystectomy should be discussed with the subject as part of the informed consent process.
* Ineligibility factors for radical cystectomy may include, but are not limited to:
* Cardiovascular disease (e.g., recent acute coronary syndrome, arrhythmia, heart failure)
* Chronic obstructive pulmonary disease that would preclude a safe surgical procedure, as determined by the treating surgeon
* Poor performance status
* Prior major abdominal and pelvic surgery that would preclude a safe surgical procedure, as determined by the treating surgeon

Cohort C Only:

* Are willing to undergo a standard of care examination under anesthesia or cystoscopy within four weeks of scheduled radical cystetomy.
* In subjects previously treated with pembrolizumab for BCG-unresponsive NMIBC that are found to have disease persistence, the disease persistence must have been confirmed no earlier than 12 weeks after initiation of pembrolizumab; subjects previously treated with pembrolizumab that are found to have disease recurrence or progression from HG Ta and/or CIS to T1 disease prior to 12 weeks after initiation of pembrolizumab may be included after discussion with the Principal Investigator.
* Patients who have received prior cisplatin-based neoadjuvant chemotherapy may be included in the study
* Age ≥18 years on day of signing informed consent.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤2 / Karnofsky performance status ≥60%, as assessed within 28 days prior to treatment initiation.
* Required values for screening laboratory tests, performed within 28 days prior to treatment initiation:

Absolute neutrophil count (ANC) ≥1000/mm3

* Platelets >75,000/mm3 without
* Hemoglobin >8 g/dL
* Creatinine clearance >40 mL/min for the dose-escalation phases, >25 mL/min for the dose expansion phases (estimated GFR can also be used in place of creatinine clearance)
* AST/ALT ≤3 times the institutional upper limit of normal (ULN)
* Total bilirubin ≤1.5 times the institutional ULN

  * Female subjects of childbearing potential must have a negative serum pregnancy test within 72 hours prior to receiving the first dose of study treatment.
  * Female subjects will be considered of non-reproductive potential if any of the following:
  * Postmenopausal [defined as at least 12 months with no menses without an alternative medical cause; in women <45 years of age a high follicle stimulating hormone (FSH) level in the post-menopausal range may be used to confirm a post-menopausal state in women not using hormonal contraception or hormonal replacement therapy. In the absence of 12 months of amenorrhea, a single FSH measurement is insufficient.
  * Have had a hysterectomy and/or bilateral oophorectomy, bilateral salpingectomy, or bilateral tubal ligation/occlusion, at least 6 weeks prior to screening
  * Has a congenital or acquired condition that prevents childbearing
  * Male and female subjects of childbearing potential must agree, if participating in sexual activity that could lead to pregnancy, to use of an adequate method of contraception from the day of study medication initiation (or 14 days prior to the initiation of study medication for oral contraception) throughout the study period up to 120 days after the last dose of trial therapy. Subjects should be informed that taking the study medication(s) may involve unknown risks to the fetus (unborn baby) if pregnancy were to occur during the study.

Male subjects will be considered of non-reproductive potential if they have azoospermia (whether due to vasectomy or an underlying medical condition). Female subjects will be considered of non-reproductive potential if as described above. Acceptable methods of contraception:

* Single method (one of the following is acceptable): intrauterine device, vasectomy of a female subject's male partner, or contraceptive rod implanted into the skin
* Combination method (requires use of two of the following): diaphragm with spermicide (cannot be used in conjunction with cervical cap/spermicide), cervical cap with spermicide (nulliparous women only), contraceptive sponge (nulliparous women only), male condom or female condom (cannot be used together), or hormonal contraceptive [oral contraceptive pill (estrogen/progestin pill or progestin-only pill), contraceptive skin patch, vaginal contraceptive ring, or subcutaneous contraceptive injection
* Male subjects must agree not to donate sperm during and after the study
* Able to comply with the treatment schedule as determined by the participant and the licensed practitioner.

Exclusion Criteria:

(Cohort A and B)

* History of or currently being treated for muscle-invasive (T2, T3, T4) locally-advanced non-resectable or metastatic urothelial carcinoma.
* Evidence of concurrent extravesical (i.e., urethra, ureter, or renal pelvis) urothelial cell carcinoma.
* Concurrent anti-cancer therapy, including investigational agents

Exceptions include:

* Cohorts A and B Exceptions: Subjects on topical therapy (e.g. topical 5-
* Cohort C Exceptions: Subjects on topical therapy (e.g. topical 5-fluorouracil) and Neoadjuvant chemotherapy (e.g. cisplatin and gemcitabine)
* Has undergone any intervening intravesical chemotherapy or immunotherapy from the time of most recent cystoscopy/TURBT to starting trial treatment (a single dose of intravesical treatment given as part of the most recent cystoscopy/TURBT, during the screening period, such as with chemotherapy as per local/regional practices, is acceptable).
* Has had prior chemotherapy, targeted small molecule therapy, cytokine therapy, or radiation therapy within 2 weeks prior to the first dose of trial treatment or who has not recovered (i.e., Grade ≤1 or at baseline) from AEs due to a previously administered agent.

  °Subjects with Grade ≤2 neuropathy or Grade ≤2 alopecia are an exception to this criterion and may qualify for the study
* Major surgery or a wound that has not fully healed within 4 weeks prior to the first dose of trial treatment.

  ° If subject has undergone major surgery greater than 4 weeks prior, subject must have recovered adequately from the toxicity and/or complications from the intervention prior to starting trial therapy
* Known additional malignancy that has had progression or has required active treatment in the last three years

Exceptions include:

* Basal cell carcinoma of the skin
* Squamous cell carcinoma of the skin that has undergone potentially curative therapy
* In situ cervical cancer
* History of prostate cancer treated with definitive intent (surgical or radiation therapy), provided that the following criteria are met: stage T2N0M0 or lower with a Gleason score ≤7 and prostate-specific antigen (PSA) undetectable for at least 1 year while off androgen deprivation therapy, that was either treated with definitive intent or untreated in active surveillance that has been stable for the past year prior to study enrollment

  * Active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease-modifying agents, corticosteroids, or immunosuppressive agents). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
  * Diagnosis of immunodeficiency, concurrent immune suppressive disease, or is receiving systemic corticosteroid therapy or any other form of immunosuppressive therapy within 4 weeks prior to the planned first dose of trial treatment. The use of physiologic doses of corticosteroids as replacement therapy (for adrenal or pituitary insufficiency, etc.) is acceptable. Topical and inhaled corticosteroids in standard doses are acceptable.
  * Known contraindications to intravesical therapy:
* Febrile illness, symptomatic urinary tract infection, or persistent gross hematuria
* Traumatic catheterization or gross hematuria on day of treatment

  * Active infection requiring systemic therapy, including active or intractable urinary tract infection within 4 weeks prior to the first dose of trial treatment
  * Severe infection within 4 weeks prior to the first dose of trial treatment, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia.
  * History of (non-infectious) pneumonitis that required steroids or current pneumonitis.
  * History of Human Immunodeficiency Virus (HIV) infection (e.g., positive HIV-1/2 antibodies).
  * Active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C [e.g., HCV RNA (qualitative) detected] infection; subjects with past/resolved Hepatitis B Virus (HBV) infection (defined as having a negative HBsAg and a positive antibody to Hepatitis B core antigen) or Hepatitis C Virus (HCV) infection are eligible only if polymerase chain reaction (PCR) testing is negative for HBV DNA or HCV RNA, respectively (must be obtained within 28 days prior to treatment initiation).
  * Pregnant or breastfeeding, or expecting to conceive within the projected duration of the trial, starting with the screening visit through 120 days after the last dose of trial treatment
  * History of stroke or intracranial hemorrhage within 6 months prior to enrollment.
  * History of pulmonary embolism or any other thromboembolic event within 6 months prior to enrollment.
  * History of undergoing an allogeneic tissue/solid organ transplant
  * History or current evidence of any condition, therapy, or laboratory abnormality that might interfere with the subject's participation for the full duration of the trial, interfere with the subject's ability to cooperate with the requirements of the trial, confound the results of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2021-11-08 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
MTD/RP2D (Cohort A) | 2 years
  The MTD will be defined as the dose level at which the estimated DLT rate from the MCRM model is closest to the target acceptable rate of 20%. If an MTD is not found after the full dose escalation study has been completed, the next dose recommended by the MCRM algorithm will be considered the RP2D. A DLT will be defined as the occurrence of any clinically significant grade 3 or 4 AE (per CTCAE version 5.0) within the DLT evaluation period that is considered by the Principal Investigator or designee to be possibly, probably, or definitely related to 2141-V11.
Reported number of adverse events from baseline (start of 2141-V11 administration) up until the last follow-up visit after 2141-V11 administration (Cohort B) | 1 year
  AE severity should be graded using CTCAE version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Bochner, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm